CLINICAL TRIAL: NCT04483713
Title: Evidence-Based Practice: Proposed Application of Facilitating Tools for Clinical Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EBP nursing Brazil
Record Dates: First submitted 2020-07-06; First posted 2020-07-23 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2021-02

CONDITIONS: Evidence-Based Practice
Keywords: Evidence-Based Practice; Evidence-Based Nursing; Education; Nursing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational Workshop (Active Comparator): Will receive theoretical and practical training in EBP through a workshop in a structured model with themes related to the introduction to EBP, with the final proposal of a practical class that aims to structure and describe an individual case through an exercise formulated to go through the phases of a project of EBP, to base this exercise we will use a finished and consolidated project, this will be used as a template of the exercise, the description of this exercise is in the programmatic content.
  Interventions: Behavioral: Educational Workshop
- Educational Workshop plus J. H. N. EBP Guide Tools (Active Comparator): Will receive the same training as group "Educational Workshop", plus the presentation and availability of the Johns Hopkins Nursing Evidence-based Practice guide tools to be used in the practice class for the structuring and individual description of the EBP exercise case. The same theme of the case will be used in both groups.
  Interventions: Behavioral: Educational Workshop; Behavioral: Educational Workshop plus J. H. N. EBP Guide Tools

INTERVENTIONS:
Behavioral: Educational Workshop — The workshop proposes a review of all stages of EBP which includes approaches to clinical care based on science and the quality of evidence, with the ultimate goal of promoting safe and quality care.
  The workshops comprise one for each group with a total workload of six (6) hours divided into two days, lasting three hours each day. The first day will be a theoretical approach and the second day a practical approach.
  The workshops with theoretical content and practical classes will be held in rooms of Albert Einstein Hospital.
  All participants of both educational strategies will answer the same questionnaires.
Behavioral: Educational Workshop plus J. H. N. EBP Guide Tools — In addition to the workshop. It will follow the same molds as the case of group "Educational Workshop" plus the Johns Hopkins Nursing Evidence-based Practice guide tools since the beginning of this practical class, when the participant will receive a description of a problem as a basis for elaborating their clinical question, and thus, move on to the next stage.
  The tools will be offered in the case of this group: question development, evidence level and quality guide, research evidence assessment tool, individual evidence tool, evidence synthesis and recommendation tool, action planning tool and tool dissemination.
  Arms: Educational Workshop plus J. H. N. EBP Guide Tools

SUMMARY:
Randomized study of educational intervention, comparative and prospective about Evidence Based Practice (EBP) and its application by clinical nurses in the implementation of EBP projects in search of best practice in nursing processes.

DETAILED DESCRIPTION:
Evidence Based Practice (EBP) has become an important issue in nursing. It is considered a process consisting of sequential steps. Multiple barriers are found, among them, time restriction, lack of personal motivation, professional resistance to research and inadequate knowledge. The proposal of this study is to provide Brazilian clinical nurses with tools to be used as a guide, with a structured process in stages as a facilitator of the implementation of EBP projects in search of best practice in nursing processes, for this the investigators will verify the adequacy of authorized translation of the Portuguese version of the Johns Hopkins Center for Evidence-Based Practice guide tools and whether these tools are facilitators in structuring and describing an EBP project from the perspective of the clinical nurse, in addition to verifying whether the EBP project met the requirements of preparation from the perspective of the researcher.

ELIGIBILITY:
Inclusion Criteria:

* Clinical nurse with a minimum of two years of training in nursing undergraduate
* Self-referred intermediate English for reading

Exclusion Criteria:

-Have previously participated in an EBP project, EBP council or research project, or have a master's or doctor's degree.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2020-12-13 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Questionnaire to check the suitability of the authorized translation of the portuguese language version of the johns hopkins evidence-based practice guide tools. | Change from Baseline suitability of the translation of the portuguese language version of the johns hopkins PBE guide tools at immediate post this intervention, an average of 3 months.
  The questionnaire have closed-ended question about the intelligibility of translation for experts, with the possibility of answering yes or no, and an open field for suggestions for changes. In case of inadequacy (which we define as less than four yes answers for the tools), we will make the changes cited by the experts and submit the changed tools to a further expert evaluation.
Questionnaire for the evaluation of the structuring process and description of an evidence-based practice project, from the perspective of the clinical nurse. | Change from Baseline evaluation of the structuring process and description of an evidence-based practice project, from the perspective of the clinical nurse, at immediate post intervention, through study completion, an average 1 year.
  The instrument has seven questions and one open for comments. The closed questions are related to the description of a clinical question with answer possibilities (very slow; slow; fast; very fast), ease in searching for evidence (challenging; difficult; easy; very easy), understanding of scientific articles (not understandable; partially understandable; understandable; totally understandable), ease in summarizing and classifying the levels of evidence and ease in describing the application of evidence with (challenging; difficult; easy; very easy), elaborating an action plan for disseminating the evidence, in addition to the ease of going through all the phases of a PBE project in relation to the material offered during the workshop (with or without Johns Hopkins tools) with answer possibilities (not helpful; partially helpful; helpful; very helpful), the latter responses are associated with greater ease in the process of structuring and describing an evidence-based practice project.
Compliance verification questionnaire in the exercise of preparing a PBE project, from the researcher's perspective. | Change from Baseline Compliance verification in the exercise of preparing a PBE project, from the researcher's perspective, at immediate post intervention, through study completion, an average 1 year.
  This tool have five closed questions to verify compliance with the basic requirements and key elements of an EBP project. The closed questions are related to the description of a clinical question with answer possibilities (yes; no), about survey of bibliographic articles with answer possibilities (Sufficient; Partially sufficient; Insufficient), about the classification of evidence according to the level of quality, elaboration of synthesis of the findings relating to the levels of evidence and ability to develop a dissemination plan for the implementation of the PBE project , with answer possibilities ( Yes; Partially; No). The latter answers are associated with a poor conformity in the exercise of structuring and describing an evidence-based practice project from the researcher's perspective.

SECONDARY OUTCOMES:
Evidence-Based Practice Questionnaire (EBPQ) | Change from de Baseline Evidence-Based Practice at immediate post intervention, through study completion, an average 1 year.
  It is a self-applicable instrument, considered important for assessing the use, opinions and knowledge of nurses about this practice. The instrument assesses attitudes, knowledge and implementation of PBE, uses a Likert-type scale with a score from one, just like never to seven equal to often, in three domains: practice, attitudes and knowledge related to PBE, with higher scores indicating more positive attitudes toward EBP.

CONTACTS AND LOCATIONS:
Overall Officials: Eliseth R Leão, PhD, Principal Investigator — Hospital Israelita Albert Einstein - Research Institute
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, Brazil

REFERENCES:
- [Background] Pereira F, Salvi M, Verloo H. Beliefs, Knowledge, Implementation, and Integration of Evidence-Based Practice Among Primary Health Care Providers: Protocol for a Scoping Review. JMIR Res Protoc. 2017 Aug 1;6(8):e148. doi: 10.2196/resprot.7727. PMID 28765102
- [Background] Friesen-Storms JH, Moser A, van der Loo S, Beurskens AJ, Bours GJ. Systematic implementation of evidence-based practice in a clinical nursing setting: a participatory action research project. J Clin Nurs. 2015 Jan;24(1-2):57-68. doi: 10.1111/jocn.12697. Epub 2014 Sep 25. PMID 25258116
- [Background] Danski MTR OG, Pedrolo E, Lind J, Johann D. A Importância da Prática Baseada em Evidências nos Processos de Trabalho do Enfermeiro. Cienc Cuid Saude 2017 Abr-Jun; 16(2). 2017
- [Background] Schneider LR, Pereira RPG, Ferraz L. A prática baseada em evidência no contexto da Atenção Primária à Saúde. Saúde debate. 2018;42(118):594-605
- [Background] Warren JI, McLaughlin M, Bardsley J, Eich J, Esche CA, Kropkowski L, Risch S. The Strengths and Challenges of Implementing EBP in Healthcare Systems. Worldviews Evid Based Nurs. 2016 Feb;13(1):15-24. doi: 10.1111/wvn.12149. PMID 26873372
- [Background] Pintz C, Zhou QP, McLaughlin MK, Kelly KP, Guzzetta CE. National Study of Nursing Research Characteristics at Magnet(R)-Designated Hospitals. J Nurs Adm. 2018 May;48(5):247-258. doi: 10.1097/NNA.0000000000000609. PMID 29629911
- [Background] Wilson M, Sleutel M, Newcomb P, Behan D, Walsh J, Wells JN, Baldwin KM. Empowering nurses with evidence-based practice environments: surveying Magnet(R), Pathway to Excellence(R), and non-magnet facilities in one healthcare system. Worldviews Evid Based Nurs. 2015 Feb;12(1):12-21. doi: 10.1111/wvn.12077. Epub 2015 Jan 16. PMID 25598144
- [Background] Magnet Recognition Program [homepage na internet]. ANCC Magnet Recognition Program® [acesso em 15/09/2019]. https://www.nursingworld.org/organizational-programs/magnet/.
- [Background] Leão ER, Farah OG, Reis EAA, Barros CGd, Mizoi CS. Perfil acadêmico, crenças e autoeficácia em pesquisa de enfermeiros clínicos: implicações para o Programa de Pesquisa de Enfermagem de um Hospital na Jornada Magnet®. Einstein (São Paulo). 2013;11(4):507-13
- [Background] Camargo FC IH, Pereira GA, Souza RM, Garcia LAA, Monteiro DAT et al. . Estratégias para o ensino da prática baseada em evidências na formação de enfermeiros: Revisão Intergrativa. REFACS (online) 2018; 6(Supl 1):363-374.
- [Background] Camargo FC PG, Iwamoto HH, Lorena LT, Goulart MB, Contim B. Oficinas para o desenvolvimento da prática baseada em evidências entre lideranças de enfermagem: estudo piloto. Rev Eletr Enf [Internet]. 2017;19:a50
- [Background] Ashktorab T, Pashaeypoor S, Rassouli M, Alavi-Majd H. Nursing Students' Competencies in Evidence-Based Practice and Its Related Factors. Nurs Midwifery Stud. 2015 Dec;4(4):e23047. doi: 10.17795/nmsjournal23047. Epub 2015 Dec 1. PMID 26835462
- [Background] Kim JS, Gu MO, Chang H. Effects of an evidence-based practice education program using multifaceted interventions: a quasi-experimental study with undergraduate nursing students. BMC Med Educ. 2019 Mar 4;19(1):71. doi: 10.1186/s12909-019-1501-6. PMID 30832639
- [Background] Camargo FC, Iwamoto HH, Galvao CM, Pereira GA, Andrade RB, Masso GC. Competences and Barriers for the Evidence-Based Practice in Nursing: an integrative review. Rev Bras Enferm. 2018 Jul-Aug;71(4):2030-2038. doi: 10.1590/0034-7167-2016-0617. English, Portuguese. PMID 30156693
- [Background] Schaffer MA, Sandau KE, Diedrick L. Evidence-based practice models for organizational change: overview and practical applications. J Adv Nurs. 2013 May;69(5):1197-209. doi: 10.1111/j.1365-2648.2012.06122.x. Epub 2012 Aug 9. PMID 22882410
- [Background] Camargo FC, Iwamoto HH, Galvão CM, Monteiro DAT, Goulart MB, Garcia LAA. Modelos para a implementação da prática baseada em evidências na enfermagem hospitalar. Texto contexto - enferm. 2018;26(4).
- [Background] Center for Evidence-Based Practice [homepage na internet]. Johns Hopkins Medicine [acesso em 07/11/2019]. Disponível em: https://www.hopkinsmedicine.org/evidence-based-practice/ijhn_2017_ebp.html
- [Background] Triolo PK, Scherer EM, Floyd JM. Evaluation of the Magnet Recognition Program. J Nurs Adm. 2006 Jan;36(1):42-8. doi: 10.1097/00005110-200601000-00010. PMID 16404200
- [Background] BARROS CGL, E. R. ; REIS, E. A. A. ; FARAH, O. G. . Excelência Assistencial: a Designação Magnet. Prática Hospitalar. 2012:São Paulo, p. 59 - 63.
- [Background] McClure ML. Magnet hospitals: insights and issues. Nurs Adm Q. 2005 Jul-Sep;29(3):198-201. doi: 10.1097/00006216-200507000-00003. PMID 16056153
- [Background] Aiken LH, Poghosyan L. Evaluation of "magnet journey to nursing excellence program" in Russia and Armenia. J Nurs Scholarsh. 2009;41(2):166-74. doi: 10.1111/j.1547-5069.2009.01268.x. PMID 19538701
- [Background] Barton SJ, Forster EK, Stuart ME, Patton AM, Rim JS, Torowicz DL. New knowledge, innovations, and improvement in a Magnet(R) Children's Hospital Cardiac Center. J Pediatr Nurs. 2012 Jun;27(3):271-4. doi: 10.1016/j.pedn.2011.07.002. Epub 2011 Sep 6. PMID 22525816
- [Background] Tinkham MR. The road to magnet: implementing new knowledge, innovations, and improvements. AORN J. 2013 May;97(5):579-81. doi: 10.1016/j.aorn.2013.02.004. No abstract available. PMID 23622830
- [Background] Delors J. Learning: the treasure within; report to UNESCO of the International Commission on Education for the Twenty-first Century (highlights)2010
- [Background] Rospendowiski K, Alexandre NMC, Cornélio ME. Cultural adaptation to Brazil and psychometric performance of the "Evidence-Based Practice Questionnaire". Acta paul enferm. 2014;27(5):405-11
- [Background] Joint Commission International. Joint Commission International survey process guide for clinical care program certification. 3ª Edição, 2014

DOCUMENTS (2):
  • Study Protocol (2019-11-11): https://cdn.clinicaltrials.gov/large-docs/13/NCT04483713/Prot_000.pdf
  • Informed Consent Form (2020-01-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT04483713/ICF_001.pdf